CLINICAL TRIAL: NCT03443232
Title: The Effect of Cryoballoon and Radiofrequency Ablations on Left Atrial Structural and Electrical Remodeling in Patients With Drug-refractory Persistent Atrial Fibrillation
Brief Title: Effect of Catheter Ablation on Left Atrial Function in Persistent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, xieruiqin, director of cardiology department, The Second Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: xierqdoctorAF
Record Dates: First submitted 2018-02-07; First posted 2018-02-23 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoballoon ablation group (Experimental): Persistens atrial fibrillation in Cryoballoon ablation group will apply cryoablation
  Interventions: Procedure: Cryoballoon ablation
- Radiofrequency ablation group (Other): Persistens atrial fibrillation in Radiofrequency ablation group will apply Radiofrequency ablation
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Cryoballoon ablation — Cryoablation is performed using a single cryoballoon.In general, the cryoablation of each pulmonary vein is carried out twice. According to the objective condition, the operator determine whether or not to carry out an additional cryoablation. Then we will applicate electrophysiological substrate mapping for guiding ablation of atrial fibrillation,If mapping system detect a poor substrate,we should continue to ablate for left atrial roof and posterior line.
  Arms: Cryoballoon ablation group
Procedure: Radiofrequency ablation — Each patient randomly allocated into the radiofrequency ablation group receives circumferential pulmonary vein isolation(CPVI),The default strategy is to create a circle surrounding the two ipsilateral pulmonary veins.We will mapping the left atrial subtrate. If mapping system detect a poor substrate,we should continue to ablate for left atrial roof and posterior line.
  Arms: Radiofrequency ablation group

SUMMARY:
A total of 106 patients with drug-refractory persistent atrial fibrillation, who are planned to undergo circumferential pulmonary vein isolation (CPVI), will be randomly allocated into two groups. These patients will receive cryoballoon ablation, radiofrequency ablation under the guidance of 3D mapping respectively (allocation ratio, 1:1). Atrial electrical activity including atrial effective refractory period, atrial conduction time, electromechanical conduction time, P wave dispersion and spatial dispersion of atrial refractory will be measured before and after the operation. Left atrial appendage flow velocity of all patients are measured by Transesophageal Echocardiography(TEE) 24 hours before the operation. Real-time ultrasound examinations of left atrial function are carried out for all patients before the operation and after the operation. Blood samples are extracted in all patients before the operation and after the operation.This study will clarify whether these different operation methods have different effects on the recovery of postoperative left atrial function and electrical activity in patients with persistent atrial fibrillation, and whether changes in left atrial function electrical activity are related to indicators such as inflammation, blood clotting and myocardial injury. Cryoballoons ablation is still less used to operate on persistent atrial fibrillation. To investigate the ablative effect, electrical remodeling and structural remodeling of persist atrial fibrillation with different operating methods. Therefore, the ablation is related indicators such as the success rate of the operation, intraoperative complications, postoperative recurrence rate and the amount of x-ray exposure are compared among two groups. At the same time, biochemical indicators of inflammation, blood clotting and myocardial injury such as blood routine, myocardial enzyme, BNP, troponin I and D-D dimmer are detected to analyze and determine which indicators are related to the postoperative recurrence of atrial fibrillation, the recovery of postoperative left atrial function.

DETAILED DESCRIPTION:
From February 2018 to February 2020, the investigators enroll consecutive patients with drug-refractory persistent atrial fibrillation who were scheduled for an initial catheter ablation.Patients are divided in to two group: persistent AF in radiofrequency ablation group, cryoballoon ablation group.

1. Radiofrequency ablation group: Each patient randomly allocated into the radiofrequency ablation group receives circumferential pulmonary vein isolation(CPVI), if atrial flutter is diagnosed before and during operation,then a radiofrequency is used to ablate cavo-tricuspid isthmus. Under the 3D electro-anatomical mapping system (Carto 3, Biosense Webster), after passing through the transseptal sheath, the ablation catheter is infused under pressure to enter into the left atrium to carry out radiofrequency ablation.The default strategy is to create a circle surrounding the two ipsilateral pulmonary veins. The cardioversion is performed if spontaneous conversion is not observed after CPVI. Observation is carried out for 20-30 minutes after the entrance and exit block of pulmonary vein potentials,in the meantime investigators will mapping the left atrial substrate. If mapping system detect a poor substrate,the investigators should continue to ablate for left atrial roof and posterior line.The situation of pulmonary vein potential conduction will be detected again. If there is a recovery, ablation will be continuously carried out.
2. Cryoballoon ablation group: Cryoablation is performed using a single cryoballoon. The diameter of the cryoballoon (Arctic Front Advance™ Cardiac CryoAblation Catheter; Medtronic, Minneapolis, MN) is determined as 28 mm or 23 mm according to pulmonary venography results. After passing through the transseptal sheath, the cryoballoon catheter enters into the left atrium and is continuously infused with heparin saline through a 15F oriented sheath. The balloon is inflated at the entrance of the pulmonary vein. The mapping confirms that the balloon blocks the entrance of the pulmonary vein. After blocking of the entrance of the pulmonary vein is enhanced, liquid nitrogen is injected for cryoablation. Before performing right pulmonary vein ablation, a secondary catheter is placed into the superior vena cava during the cryoablation. A cycle length of 999 ms is taken to continuously make the right phrenic nerve pulsate. If diaphragm movement is weakened or disappears, the cryoablation will be immediately stopped. In general, the cryoablation of each pulmonary vein is carried out twice. According to the objective condition, the operator determine whether or not to carry out an additional cryoablation. The cardioversion is performed if spontaneous conversion is not observed after CPVI. Then investigators will applicate electrophysiological substrate mapping for guiding ablation of atrial fibrillation,If mapping system detect a poor substrate, investigators should continue to ablate for left atrial roof and posterior line. By testing the entrance and exit block of pulmonary vein potentials，the investigators observe the duration of potentials.
3. All patients fill the follow-up form before operation. After catheter ablation therapy, all patients invited to come back to the outpatient clinic every week in the first month, and then at 2, 3, 6, 9, and 12 month to follow up. Patients received electrocardiogram and Holter monitor examination if with symptoms of palpitations. Those patients with no symptoms received electrocardiogram every month and Holter monitor examination every 6 months. Recurrence of atrial fibrillation was defined as atrial fibrillation/flutter or atrial tachycardia lasting ≥ 30 seconds 3 months after ablation therapy. Atrial electrical activity including atrial effective refractory period, atrial conduction time, electromechanical conduction time, P wave dispersion and spatial dispersion of atrial refractory will be measured before and after the operation.Blood samples (routine blood, high sensitivity c-reactive protein,B-type natriuretic peptide (BNP), cystatin C,homocysteine,β2-microglobulin) and transthoracic echocardiography indexes (left atrial anterior to posterior diameter, left atrial length-diameter,left atrial transverse-diameter,left atrial volume index, mitral e', E peak, A peak, E/A,velocity time integral (VTI), left atrial ejection fraction, left atrial strain, strain rate and atrial electrical - mechanical conduction time) are recorded in all patients at each follow-up. Patients with AF recurrence must have an electrocardiogram or a 24 hour holter monitor evidence.

ELIGIBILITY:
Inclusion Criteria:Persistent

* Persistent AF is defined as AF that persists without interruption for 7 days (electrocardiogram data or Holter), atrial fibrillation cannot be prevented in patients who orally take class I and III antiarrhythmic drugs, and patient age is <80 years.

Exclusion Criteria:

* •left ventricular dysfunction

  * atrial thrombosis
  * valvular heart disease
  * hyperthyroidism
  * patients who underwent prosthetic heart valve replacement
  * patients with previous history of atrial fibrillation ablation
  * pregnant women
  * patients with existing liver and kidney disease
  * malignant tumors
  * hematological system diseases

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Change of P wave | 1-12 month
  Electrocardiogram
Atrial electrical activity | During the operation
  Electrophysiological examination
Left atrial function of postoperative | 1-12 month
  Transthoracic echocardiography

SECONDARY OUTCOMES:
Plasma biomarkers of inflammation assessed | 1-12 month
  Blood samples are extracted in all patients to detected
B type natriuretic peptide assessed | 1-12 month
  Blood samples are extracted in all patients to detected
Coagulation index assessed | 1-6 month
  Blood samples are extracted in all patients to detected

OTHER OUTCOMES:
homocysteine assessed | 1-12 month
  Blood samples are extracted in all patients to detected
β2-microglobulin assessed | 1-12 month
  Blood samples are extracted in all patients to detected

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China